CLINICAL TRIAL: NCT03627351
Title: Taste of Medicines for Children: Genetic Variation and Medical Adherence (Aim 1)
Brief Title: Sensory Evaluation of the Taste of Pediatric Medicines
Acronym: MEDTASTE
Status: Completed | Type: Observational
Sponsor: Monell Chemical Senses Center (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: T24653; R01DC011287 (NIH)
Record Dates: First submitted 2018-07-09; First posted 2018-08-13 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: Taste; Odor; Sensory Panel; Flavor; Genes; Pediatric Medicines

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Identification of genetic polymorphisms in DNA from saliva samples collected at baseline that are associated with variation in flavor and palatability ratings of pediatric medicines through genome wide association study of adult panelists
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Women and Men: Group of healthy women and men

SUMMARY:
The investigators will conduct a systematic study of the sensory perception of a diverse set of commonly used pediatric liquid medications and excipients in tandem with an equally complete genetic analysis of the adult sensory panelists to investigate the relationship between genetic variation and individual differences in the perceived flavor (taste, smell, irritation) of pediatric medicines. The flavor of each medicine and excipient will be measured individually using both cognitively demanding methods unsuitable for young children and simpler measures validated for use by children. Salivary DNA samples will be collected to carry out genome wide association study (GWAS).

DETAILED DESCRIPTION:
This is a single-site, cross-sectional, repeated measures study of healthy adult panelists which will investigate individual differences in the taste of a diverse set of commonly used pediatric liquid medications (e.g., clindamycin, prednisone, dexamethasone, mercaptopurine, ibuprofen, lopinavir/ritonavir, propylthiouracil) and excipients (e.g., sucrose, citric acid, bitter agents, salt, menthol and other odors) in tandem with genetic analysis. Because the medication given to pediatric patients is the whole liquid formulation (API + excipients), the investigators' approach will be to have panelists taste (without swallowing) what patients taste. Using validated psychophysical tools such as the general labelled magnitude scale (gLMS), the hedonic gLMS, and the hedonic 5-face scale, adults panelists will rate the intensity of the basic tastes, overall intensity, irritation, or palatability (hedonics) of a variety of pediatric drugs (with and without noseclips), along with generally recognized as safe (GRAS) taste and odor stimuli commonly used in basic research and/or as excipients in many liquid formulations These data will establish whether the palatability and flavor of each medicine varies among adult panelists. From these data, the investigators will determine a) whether the dislike of one medicine by a panelist predicts their dislike of another medicine in the same class or medicines with the same excipients; b) whether variation in the flavor and palatability ratings of each medicine relates to variation in genetic polymorphisms, as determined from the GWAS; and c) whether the panelists' palatability ratings of each medicine, as assessed by the simpler hedonic 5-face scale, is significantly related to hedonic gLMS ratings.

ELIGIBILITY:
Inclusion Criteria:

- Men and women who are between the ages of 18 and 55 years

Exclusion Criteria include the following:

* For all female participants, a urine pregnancy test will be done on each testing day. Only those with a negative pregnancy test will be allowed to participate in taste testing.
* Smokers will be excluded since it alters flavor perception.
* Potential subjects will be excluded if they are on drugs with potential serious adverse effects that are mediated through CYP450 3A4 since ritonavir is a potent inhibitor of CYP450 3A4 and could lead to elevated levels of the prohibited drugs if swallowed. The prohibited drugs include the following:
* Alfuzosin (Uroxatral; alpha-1-adrenoreceptor antagonist)
* Astemizole (Hismanal; antihistamine)
* Bepridil (Vascor; calcium channel blocker)
* Cerivastatin (Baycol; statin)
* Cisapride (Propulsid; GI motility agent)
* Dronedarone (multaq; anti-arrhythmic)
* Ergotamine (Cafergot, Ergot derivatives)
* Flecainide (Tabocor; anti-arrhythmic)
* Lovastatin (Altoprev; HMG-CoA Reductase Inhibitor)
* Lurasidone (Latuda; antipsychotic)
* Midazolam (Versed; sedative/hypnotic)
* Pimozide (Orap; antipsychotic)
* Ranolazine (Ranexa; anti-anginal)
* Simvastatin (Zocor; statin)
* Terfenadine (Seldane; antihistamine)
* Tinidazole (Tindamax; anti-parasitic)
* Trazodone (Desyrel; antidepressant/sedative)
* Triazolam (Halcion; sedative)
* Warfarin (Coumadin; blood thinner)
* Potential subjects will be excluded if they have had current (within the last 24 hours) use of sildenafil (Viagra), tadalafil (Cialis), and verdenafil (Levitra) are also exclusion criteria. These drugs can be used as needed for erectile dysfunction. They are also used as a daily treatment for pulmonary arterial hypertension. With CYP450 3A4 blockade and current use, hypotension, syncope, and prolonged erection are possible.
* Potential subjects will be excluded if they have known allergies or hypersensitivity reactions to lopinavir, ritonavir, clindamycin, prednisone, dexamethasone, ibuprofen, 6-mercaptopurine, propylthiouracil, or any of the excipients in the liquid formulations to be tested.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy men and women between the ages of 18 and 55 years
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2021-07-16 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Flavor ratings (using general labelled magnitude scale, gLMS) of pediatric medicines and excipients | Through study completion, an average of 3 years
  Flavor ratings of each pediatric medicine and excipient as assessed by the general labelled magnitude scale [gLMS]; each medicine and each excipient is rated individually; range 0 [minimum, no flavor] to 100 [maximum; strongest flavor rating]
Palatability ratings (using hedonic general labelled magnitude scale, hedonic gLMS) of the flavor of pediatric medicines and excipients | Through study completion, an average of 3 years
  Ratings of the palatabillity of the flavor of each medicine and excipient, as assessed by the hedonic general labelled magnitude scale; each medicine and each excipient is rated individually, range: -100 [minimum palatability rating] to 0 [neither like nor dislike] to 100 [maximum /strongest imaginable palatability ratings]
Detect genetic associations (GWAS) with flavor and palatability ratings of pediatric medicines | After study completion, 2021-2022
  To detect genetic associations with taste and palatability ratings phenotypes of each medicine

SECONDARY OUTCOMES:
Hedonic ratings (using 5 face scale) of the flavor of pediatric medicines | Through study completion, an average of 3 years
  Ratings of the liking of the flavor of each medicine, as assessed by the simpler, hedonic 5-face scale; each medicine is rated individually; range: 1 (minimum, greatest dislike score) to 5 (maximum; greatest liking score). Each panelist's hedonic 5-face scale rating will be correlated with the more sophisticated hedonic gLMS rating for each medicine to lay the foundation for future research in pediatric populations

CONTACTS AND LOCATIONS:
Overall Officials: Julie A. Mennella, PhD, Principal Investigator — Monell Chemical Senses Center; Elizabeth Lowenthal, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Monell Chemical Senses Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
dbGAP
Supporting Information: Study Protocol, SAP
Time Frame: 2023 and for 1 year
Access Criteria: To be developed

REFERENCES:
- [Background] Mennella JA, Mathew PS, Lowenthal ED. Use of Adult Sensory Panel to Study Individual Differences in the Palatability of a Pediatric HIV Treatment Drug. Clin Ther. 2017 Oct;39(10):2038-2048. doi: 10.1016/j.clinthera.2017.08.012. Epub 2017 Sep 18. PMID 28923290
- [Background] Mennella JA, Spector AC, Reed DR, Coldwell SE. The bad taste of medicines: overview of basic research on bitter taste. Clin Ther. 2013 Aug;35(8):1225-46. doi: 10.1016/j.clinthera.2013.06.007. Epub 2013 Jul 22. PMID 23886820
- [Background] Kalva JJ, Sims CA, Puentes LA, Snyder DJ, Bartoshuk LM. Comparison of the hedonic general Labeled Magnitude Scale with the hedonic 9-point scale. J Food Sci. 2014 Feb;79(2):S238-45. doi: 10.1111/1750-3841.12342. Epub 2014 Jan 14. PMID 24422940
- [Background] Snyder DJ, Prescott J, Bartoshuk LM. Modern psychophysics and the assessment of human oral sensation. Adv Otorhinolaryngol. 2006;63:221-241. doi: 10.1159/000093762. PMID 16733341
- [Background] Bobowski N, Mennella JA. Personal Variation in Preference for Sweetness: Effects of Age and Obesity. Child Obes. 2017 Oct;13(5):369-376. doi: 10.1089/chi.2017.0023. Epub 2017 May 12. PMID 28497993
- [Background] Bobowski N, Reed DR, Mennella JA. Variation in the TAS2R31 bitter taste receptor gene relates to liking for the nonnutritive sweetener Acesulfame-K among children and adults. Sci Rep. 2016 Dec 14;6:39135. doi: 10.1038/srep39135. PMID 27966661
- [Derived] Kan M, Saraiva LR, Hwang LD, Lowenthal ED, Himes BE, Mennella JA. Genome-wide association study of the taste and hedonic ratings of the low-calorie sweetener acesulfame potassium. Sci Rep. 2025 Jul 1;15(1):22121. doi: 10.1038/s41598-025-05739-x. PMID 40594245